CLINICAL TRIAL: NCT04298762
Title: The Effect of Peer Comparison Emails on Oncologists' Documentation of Cancer Stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anna Sinaiko, Assistant Professor of Health Economics and Policy, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: staging_documentation
Record Dates: First submitted 2020-02-11; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison Group (Placebo Comparator): Physicians in the control group did not receive peer comparison emails.
  Interventions: Other: No peer comparison email
- Intervention Group (Experimental): Physicians in the intervention group received peer comparison emails.
  Interventions: Other: Peer comparison email

INTERVENTIONS:
Other: No peer comparison email — The comparison group received no email communication on their cancer stage documentation activity.
  Arms: Comparison Group
Other: Peer comparison email — The intervention group received three separate emails with individualized data on their cancer stage documentation activity in the previous 1-3 months. The email described the number and percent of attributed patients for whom cancer stage was documented, and included a figure showing their staging documentation rate compared to their peers.
  Arms: Intervention Group

SUMMARY:
Documenting cancer stage is the most important determinant of treatment approach and survival for cancer patients. However, oncologists do not routinely document a patient's cancer stage in the structured field in electronic health records. This quality improvement pilot study evaluated the impact of sending an email to physicians at a cancer center of a large academic hospital with individualized data on their rates of cancer stage documentation using a structured field. The investigators assessed patient-level documentation and physician-level rates of staging documentation over 15 months including a three-month pre-period, a six-month pilot phase and a six-month follow-up period. The investigators also estimated staging documentation rates separately for each physician's new versus established patients.

ELIGIBILITY:
Inclusion Criteria:

* Attending physicians who had been at one of three sites of hospital between January - August 2018

Exclusion Criteria:

* Physicians treating cancer patients where American Joint Committee on Cancer (AJCC) staging modules were less clinically relevant
* Physicians with low clinical volume (<5 patients over 3 months)
* Physicians without any outpatient visits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Measuring if a patient's cancer stage was documented in a structured field in the Electronic Health Record on the date of the patient's first ambulatory care visit | 15 months
  Indicator of whether the structured field for cancer stage in the patient's electronic health record (EHR) was populated on the date of the first outpatient encounter that a patient had during the study period (1=yes, 0=no)

SECONDARY OUTCOMES:
Staging documentation rate (monthly) | 15 months
  Percentage of patients whose first outpatient encounter occurred in a given month for whom cancer stage was documented

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sinaiko, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No